CLINICAL TRIAL: NCT06492031
Title: Effectiveness and Safety of Icodextrin Peritoneal Dialysis Solution (Extraneal®) for Long Dwell Exchange in Peritoneal Dialysis in Patients With Chronic Renal Failure: a Multicenter, Ambispective Cohort, Observational, Real-world Study
Brief Title: Observational Study of the Use of Extraneal in Peritoneal Dialysis in Patients
Acronym: oSCAR
Status: Recruiting | Type: Observational
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU599284
Record Dates: First submitted 2024-06-25; First posted 2024-07-09 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Chronic Renal Failure
Keywords: Continuous ambulatory peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Icodextrin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Icodextrin (ICO) Group: Icodextrin is only intended for intraperitoneal administration and is recommended for long dwell during CAPD (i.e., recommended dwell time from 8-16 hours). Administration will be done at a rate that is comfortable for the patient, typically within 10-20 minutes.
  Interventions: Drug: Icodextrin Peritoneal Dialysis Solution
- Glucose Group: During CAPD, 2L of dialysis fluid is instilled into the peritoneal cavity and allowed to dwell for a certain period. The dwell time typically ranges from 4 to 8 hours during the day and 8 to 12 hours at night. This process is repeated 3 to 4 times a day, for 6 to 7 days a week. The frequency of solution exchanges may vary for each individual to achieve desired biochemical and solution control. Most solution exchanges utilize a 1.5% or 2.5% glucose dialysis solution. If more solution removal is required, a 4.25% glucose peritoneal dialysis solution can be used. Regular measurement of the patient's weight can be used to guide the setting of ultrafiltration volume.
  Interventions: Drug: Glucose Peritoneal Dialysis Solution

INTERVENTIONS:
Drug: Icodextrin Peritoneal Dialysis Solution — The treatment modality, treatment frequency, treatment dose, duration of dwell, and length of treatment, as determined and supervised by a prescribing physician experienced in treating ESRD with PD.
  Other Names: Extraneal
  Groups: Icodextrin (ICO) Group
Drug: Glucose Peritoneal Dialysis Solution — The treatment modality, number of daily dialysate exchanges, dialysate concentration, exchange dosage of dialysate, duration of dwell, and length of treatment for PD patients as determined by the clinician.
  Groups: Glucose Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of icodextrin and glucose peritoneal dialysis (PD) solutions for the long dwell exchange in PD patients with continuous ambulatory peritoneal dialysis (CAPD), and to describe medical resource utilization in patients with PD on icodextrin.

DETAILED DESCRIPTION:
Patients will be divided into icodextrin dialysate group (ICO group) and glucose dialysate group (glucose group).

ICO group: Patient data will be collected retrospectively and prospectively. Patients currently prescribed icodextrin will be recruited and enrolled. Data for these patients will included both retrospective historical data collection as well as a prospective collection of additional data. Within the relative look-back period (i.e., within 6 months before the launch of the study site), data will be collected from baseline (i.e., the most recent medical records prior to the first prescription of icodextrin) up to signing of the ICF. After providing informed consent, patient data will be prospectively collected for 12 months.

Additionally, any patients who are first prescribed icodextrin therapy after the launch of the study site will also be recruited and enrolled prospectively and data will be collected up to 12 months from enrollment for this group. For these patients, baseline will be defined as the most recent medical record from the time of signing the ICF to the first prescription of icodextrin.

Glucose group: Patient data will be collected retrospectively. Retrospective data will be collected up to 12 months from baseline (i.e., the most recent medical record before the index date, whereby the index date is defined as the date of the first prescription of glucose PD solutions for long dwell exchange between July 1, 2020, and December 31, 2020).

The effectiveness and safety between the 2 groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria for patients enrolled retrospectively in the ICO Group:

* Age ≥ 18 years old at first prescription of icodextrin, male or female;
* With a definite diagnosis of CRF and on maintenance PD ≥ 3 months;
* On CAPD treatment;
* Being treated with icodextrin long dwell exchange with an icodextrin prescription ≤ 6 months with essential baseline information(including age, gender, PD vintage, presence of diabetes or not, PET, and assessment of dialysis adequacy);
* Voluntarily sign the informed consent form (ICF) and be willing to complete the study visits as required by the investigator (For death cases, exemption of the informed consent will be applied with approval of the ethics committee).

Inclusion Criteria for patients enrolled prospectively in the ICO Group:

* Age ≥ 18 years old, male or female;
* Patients with a definite diagnosis of CRF and on maintenance PD ≥ 3 months;
* On CAPD treatment, with planned prescription for icodextrin;
* Voluntarily sign the ICF and be willing to complete the study visits as required by the investigator.

Exclusion Criteria for the ICO Group:

* Those with combined HD within 30 days prior to enrolment;
* History of peritonitis within 30 days prior to enrolment or presence of acute or chronic exit site infection or tunnel infection at enrolment;
* Participation in another interventional study within 30 days prior to enrolment or concurrently with this study;
* Allergy to any components of Icodextrin;
* Pregnancy or in lactation;
* Any other condition for which the investigator considers the patient to be unsuitable for participation in this study.

Inclusion Criteria for the Glucose Group:

* Age ≥ 18 years at index date, male or female;
* Those with a definitive diagnosis of CRF prior to the index date and eligible for CAPD treatment with Baxter's glucose PD solutions between July 1, 2020 and December 31, 2020;
* On maintenance PD ≥ 3 months;
* Essential baseline information(including age, gender, PD vintage, presence of diabetes or not, peritoneal transport status);
* Any prescription of Baxter's glucose PD solutions and medical records of clinical events within 1 year from baseline.

Exclusion Criteria for the Glucose Group:

* Those with combined HD within 30 days prior to the index date;
* History of peritonitis within 30 days prior to the index date or presence of acute or chronic exit site infection or tunnel infection during the index period;
* Prescription of non-Baxter PD solutions within 1 month prior to the index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in China prescribed icodextrin or glucose PD solutions for continuous ambulatory peritoneal dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 889 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of the incidence of a composite endpoint for technique failure and death | 12 months
  Technique failure is defined as:
  * Treatment transferred from PD to HD/PHD > 30 days; or
  * PHD defines as adding HD treatment at least once every 2 weeks in 30 days during PD,
  Death is specified as deaths during PD or deaths within 30 days with treatment from PD to HD/PHD

SECONDARY OUTCOMES:
Comparison of the proportion of patients with technique failure | 12 months
  Number and proportion of patients with technique failure
Comparison of the incidence of cardiovascular events | 12 months
  Cardiovascular events include acute myocardial infarction, sudden severe arrhythmia ( a trial fibrillation and arrhythmia requiring hospitalization or medication), hospitalization for heart failure, stroke, and cardiovascular death.
Comparison of the incidence of the changes in ejection fraction | 12 months
  Change of the echocardiographic values from baseline: left ventricular ejection fraction fraction (LVEF）
Comparison of all-cause deaths | 12 months
  All-cause deaths refer to the total number of deaths from any cause within the study timeframe
Comparison of medical resource utilization in terms of hospitalizations | 12 months
  Excluding hospitalizations due to medicare payments or other non-medical issues. For ICO group only
Comparison of annual exchange dosage of ICO | 12 months
  For ICO group only

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Beijing Haidian Hospital, Beijing
  - Hangzhou Hospital Of Traditional Chinese Medicine, Hangzhou
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Nanjing Drum Tower Hospital, Jiangse
  - Wuxi People's Hospital, Jiangse
  - The First People's Hospital of Kunshan, Jiangse
  - Ningbo First Hospital, Ningbo
  - Shanghai General Hospital, Shanghai
  - Renji Hospital Shanghai Jaotong University School of Medicine, Shanghai
  - The Second Affiliated Hospital of Soochow University, Suzhou

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, the Sponsor will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP).
Supporting Information: Study Protocol, SAP
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If the Sponsor agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of the Sponsor prior to the release of any data.